CLINICAL TRIAL: NCT01875575
Title: Oral Glucose in Normal-weight and Obese Volunteers
Brief Title: Oral Glucose Stimulation in Normal-weight and Obese Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EKBB 08/11
Record Dates: First submitted 2013-05-08; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Endocrine System Diseases
Keywords: glucagon-like peptide-1; peptide tyrosine tyrosine; ghrelin; stomach; small intestine; gastric emptying
MeSH Terms: conditions — Endocrine System Diseases | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose 10g (Active Comparator): 10g Glucose in 200ml tap water given orally (plus 50 mg 13C-sodium acetate)via nasogastric tube
  Interventions: Dietary Supplement: Glucose 10g
- Glucose 25g (Active Comparator): 25g Glucose in 200ml tap water given orally (plus 50 mg 13C-sodium acetate)via nasogastric tube
  Interventions: Dietary Supplement: Glucose 25g
- Placebo (Placebo Comparator): intragastric tap water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Glucose 25g
  Arms: Glucose 25g
Dietary Supplement: Glucose 10g
  Arms: Glucose 10g

SUMMARY:
The objective of this study is to examine gastric emptying and satiety hormones after oral glucose stimulation in 2 different concentrations in normal-weight and obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight subjects with a body-mass index of 19.0-24.5 or healthy obese subjects with a body-mass index of > 30
* Normal eating habits
* Age 18-40 years
* Stable body weight for at least three months

Exclusion Criteria:

* Smoking
* Substance abuse
* Regular intake of medications (except for oral contraceptives)
* Medical or psychiatric illness
* Any abnormality detected during the screening procedure
* history of gastrointestinal disorders
* food allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Effect of different oral glucose loads on secretion of satiation hormones | 240min.
  Plasma concentrations of glucose, insulin, glucagon, ghrelin, GLP-1, PYY and CCK are measured

SECONDARY OUTCOMES:
Effect of different oral glucose loads on gastric emptying | 240min.
  measured by C13 breath test

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Meyer-Gerspach AC, Cajacob L, Riva D, Herzog R, Drewe J, Beglinger C, Wolnerhanssen BK. Mechanisms Regulating Insulin Response to Intragastric Glucose in Lean and Non-Diabetic Obese Subjects: A Randomized, Double-Blind, Parallel-Group Trial. PLoS One. 2016 Mar 4;11(3):e0150803. doi: 10.1371/journal.pone.0150803. eCollection 2016. PMID 26942445